CLINICAL TRIAL: NCT00002677
Title: PHASE I STUDY OF THE ORALLY ADMINISTERED BUTYRATE PRODRUG, TRIBUTYRIN, IN PATIENTS WITH SOLID TUMORS
Brief Title: Tributyrin in Treating Patients With Refractory Prostate Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC-9421; CDR0000064322 (Registry Identifier: PDQ (Physician Data Query)); NCI-T94-0181O
Record Dates: First submitted 1999-11-01; First posted 2004-05-11 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV prostate cancer; recurrent prostate cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Drug Therapy; tributyrin

ARMS (1):
- Arm I (Experimental): Patients receive oral tributyrin every 8 hours for 3 weeks. Treatment continues every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease may receive additional courses at the discretion of the protocol chairperson. Cohorts of 3-6 patients receive escalating doses of tributyrin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: chemotherapy; Drug: tributyrin

INTERVENTIONS:
Drug: chemotherapy
Drug: tributyrin

SUMMARY:
Phase I trial to study the effectiveness of tributyrin in treating patients with refractory stage IV prostate cancer or other solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and optimum schedule of tributyrin in patients with prostate cancer or other solid tumors.

II. Determine the toxic effects of tributyrin in these patients. III. Determine the pharmacodynamics of tributyrin, including modulation of tumor markers, evaluation of clinical remission (when possible), assessment of F-reticulocytes and/or F cells, and evaluation of hemoglobin F before and after treatment, in these patients.

IV. Determine the pharmacokinetics of tributyrin, including maximum plasma concentration, terminal half-life, area under the concentration time curve, volume of distribution, and clearance of butyrate, in these patients.

V. Determine the relationship between the pharmacokinetics and toxic or therapeutic pharmacodynamic effects of butyrate in these patients.

VI. Calculate a tributyrin dose, using results from pharmacokinetic and pharmacodynamic studies, that achieves sustained butyrate concentrations capable of increasing therapeutic effects with reduced toxicity.

OUTLINE: This is a dose escalation study.

Patients receive oral tributyrin every 8 hours for 3 weeks. Treatment continues every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease may receive additional courses at the discretion of the protocol chairperson. Cohorts of 3-6 patients receive escalating doses of tributyrin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven prostate cancer or other solid tumor that is refractory to standard treatment or for which no standard therapy exists
* Patients with prostate cancer must meet the following conditions:

  * Stage D2 disease
  * Disease progression after orchiectomy or treatment with leuprolide or flutamide
  * If no prior orchiectomy, must continue leuprolide or other antiandrogen throughout study
* No CNS neoplasms or brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* Life expectancy: More than 3 months
* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 1.5 times normal
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance greater than 50 mL/min
* No concurrent medical or psychiatric condition that would preclude study
* Able to swallow numerous capsules
* Willing to participate in pharmacokinetic studies
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy (more than 8 weeks since prior carmustine, mitomycin, or other drugs with delayed toxic effects) and recovered
* No prior suramin
* At least 4 weeks since prior flutamide
* No concurrent hydrocortisone or other steroids
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1995-08 (Actual); Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Van Echo, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States